CLINICAL TRIAL: NCT02810275
Title: Effect of Folic Acid on Homocysteine Levels and Flow-mediated Dilation in HIV and HIV-HCV Coinfected Patients: a Randomized Controlled Trial
Brief Title: Folinic Acid: Supplementation and Therapy
Acronym: FAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Sandra Costa Fuchs, Full Professor, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CAAE: 00533612.8.0000.5346; GPPG-140240 (Other Grant/Funding Number: Hospital de Clinicas de Porto Alegre - FIPE); RBR-9366qc (Registry Identifier: Brazilian Clinical Trials Registry (ReBEC))
Record Dates: First submitted 2016-06-19; First posted 2016-06-22 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-09

CONDITIONS: HIV Infection; HCV Coinfection
MeSH Terms: conditions — HIV Infections | interventions — Leucovorin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folinic Acid (Experimental): Folinic acid group received 5 mg daily during four weeks
  Interventions: Drug: Folinic Acid
- Placebo (Placebo Comparator): Placebo group received a tablet daily during four weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folinic Acid — Folinic acid 5 mg, taking in the morning, daily, during four weeks
  Other Names: FA
  Arms: Folinic Acid
Drug: Placebo — Placebo capsule received 1 tablet, taking in the morning, during four weeks
  Other Names: Control
  Arms: Placebo

SUMMARY:
Patients infected by HIV or HIV-HCV coinfected have higher survival due to the use of HAART, but survival is accompanied by increased morbidity and associated cardiovascular disease (CVD). Endothelial dysfunction is an early marker of atherogenesis, acting as an intermediate in the causal pathway of CVD. Folinic acid (FA) has been shown to reduce CVD outcomes, especially among individuals with hyperhomocisteinemia.

To date, few studies provided consistent information about efficacy of pharmacological interventions that minimize damage to the vascular endothelium in patients infected by HIV or HIV-HCV coinfected. The main hypothesis of this study is that FA supplementation protects the vascular endothelium, and consequently might prevent subclinical atherosclerosis. Thus, the first step is to determine the efficacy of supplementation with FA, and to compare the effect between HIV and HIV-HCV coinfected.

DETAILED DESCRIPTION:
Study design: This was a randomized placebo-controlled trial, with blinding of health care team, participants, and investigators, in which the participants were randomly assigned in a 1:1 ratio to receive FA or placebo for four weeks.

Participants: Patients receiving care for HIV, at the outpatient clinic of the Hospital Universitario de Santa Maria, in southern Brazil, from October 2012 to September 2013, were recruited. Eligible participants: HIV infected or HIV-HCV coinfected patients, 18-50 years, men and women, receiving HAART, had undetectable viral load for more than six months. Patients were excluded: patients with diabetes mellitus, previous acute myocardial infarction, myocardial revascularization, or stroke, creatinine >1.5 mg/dL, clinical diagnosis or ultrasound, endoscopic, or laboratory evidence of liver cirrhosis, on treatment with statins, fibrates, hormone replacement therapy, sulfonamides, vitamin supplements, or FA in the last 30 days, and pregnant women.

Intervention Patients assigned to the intervention group received FA 5 mg, per oral, once a day, in the morning, during four weeks. Patients assigned to the placebo group received the same prescription. The trial provided FA and placebo in tablet form, identical in color, smell, taste, shape, and size. Both FA and placebo were prepared in a single batch, in an independent laboratory, by a pharmacist with no involvement in the trial. They were pre-packed in bottles containing 30 tablets each, individually labeled with an alphanumeric code and stored.

Outcomes The primary endpoint were changes in homocysteine, vitamin B12 levels, and brachial artery FMD during reactive hyperemia, as measured by Doppler ultrasound, from randomization to the end of follow-up. FMD was characterized by the variation in mean arterial flow measured as the peak change in vessel diameters relative to the baseline.

Sample size Sample size was calculated based on the results of a previous RCT,(14) which used plethysmography to measure FMD. To detect a difference of at least 6% between intervention and placebo groups, with standard deviations ranging from 5% to 7%, we calculated that a sample size of at least 17 patients per group, with randomization stratified by HCV coinfection status, was required to achieve 80% power and a 95% confidence interval.

ELIGIBILITY:
Inclusion criteria:

* HIV infected patients
* HIV-HCV coinfected patients
* 18-50 years
* men and women
* receiving HAART
* with undetectable viral load for more than six months.

Exclusion Criteria:

* Patients with diabetes mellitus,
* previous CVD: acute myocardial infarction, myocardial revascularization, or stroke,
* creatinine >1.5 mg/dL,
* clinical diagnosis or ultrasound, endoscopic, or laboratory evidence of liver cirrhosis,
* on treatment with: statins, fibrates, hormone replacement therapy, sulfonamides, vitamin supplements, or FA in the last 30 days,
* pregnant women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation | Four weeks
  The response was defined by the variation in the flow mediated dilatation between intervention and placebo groups.

SECONDARY OUTCOMES:
Serum homocysteine | Four weeks
  Variation in the serum homocysteine between intervention and placebo groups.

OTHER OUTCOMES:
Blood pressure | Four weeks
  The response was defined by variation in blood pressure between intervention and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra C Fuchs, PhD, MD, Study Chair — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: No